CLINICAL TRIAL: NCT01075360
Title: The Role of Aromatic Hydrocarbon Receptor in the Tumorigenesis of Neuroblastoma and Its Relationship With MYCN Expression
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Wen-Ming Hsu, National Taiwan University Hospital
Other Study IDs: 200806005R
Record Dates: First submitted 2010-02-23; First posted 2010-02-25 (Estimated); Last update posted 2010-02-25 (Estimated); Status verified 2010-02

CONDITIONS: Neuroblastoma
Keywords: Neuroblastoma, MYCN, AHR
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Neuroblastoma (NB) is the most common malignant tumor of infancy. Approximately 60% of NB patients are clinically diagnosed as the stage IV disease and have a very poor prognosis with the 5-year survival rate no more than 30%. Molecular markers of NB have great impacts on the tumor behavior. MYCN amplification is the most well-known marker to predict a poor outcome in NB patients. However, how MYCN affects the NB cell behavior remains unknown. In our preliminary studies, we performed a genome-wide analysis of the differential gene expression in 10 NB tumors with MYCN amplification and 10 with normal MYCN copy number. We found that aromatic hydrocarbon receptor (AHR) reversely correlated with the MYCN expression. This relationship was verified in 83 NB tumor samples. In addition, positive AHR expression by immunostaining of NB tumors predicted a favorable prognosis. These lines of evidence demonstrate that AHR not only relates to the MYCN expression but also plays an important role in the tumorigenesis of NB. Therefore in this project we aim at further studying the relationship between AHR and MYCN. In addition, the possible role of AHR in the tumorigenesis of NB will be clarified. Specifically, we propose a 3-year project with the following three aims:

Aim I. Determine the molecular relationship between AHR and MYCN expression. AHR has been shown to suppress the E2F1 expression. E2F1 reversely has been found to upregulate the expression of MYCN. In our preliminary microarray study, we also found that the expression E2F1 positively correlated with the MYCN expression but inversely correlated with the expression of AHR. Therefore, NB cells will be transfected with AHR expression vector or AHR siRNA, then the associated E2F1 and MYCN expression will be examined to clarify if AHR could regulate MYCN expression via E2F1. Furthermore, the E2F1 levels will also be manipulated to determine if the effect of AHR on MYCN depends on E2F1. In addition, the E2F1 expression in NB tumor samples will also be examined to clarify its in vivo role.

Aim II. Determine the effect of AHR expression on the NB cell behavior. The baseline AHR expression levels in several NB cell lines will be examined. AHR is then overexpressed by gene transfection in NB cells. The cell proliferation, migration, and differentiation after AHR overexpression are evaluated. Furthermore the AHR expression in normal neuron cells is also examined, and suppressed by siRNA to if downregulation of AHR could lead to cancer development.

Aim III. Determine if AHR could be a target of gene therapy for NB. NB cells with either normal MYCN or MYCN amplification before and after AHR gene transfection are inoculated into nude mice to demonstrate the effect of AHR expression on NB cells behavior in vivo. AHR is then transfected into the wild type NB tumor to see if the tumor growth could be suppressed by AHR expression. Then wild type tumor and tumors transfected with AHR are subjected microarray analysis to compare with the human tumor data set for evaluation of gene expression changes along with differential AHR expression. Altogether, our studies will not only establish the relationship between AHR and MYCN, but also allow us to depict the functional role of AHR-MYCN interaction in the tumorigenesis of NB.

ELIGIBILITY:
Inclusion Criteria:

* Neuroblastoma patients with complete follow-up and sufficient samples for study

Exclusion Criteria:

* Neuroblastoma patients without complete follow-up or sufficient samples for study

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: From year 1990 to 2009, pediatric neuroblastoma patients treated at National University Hospital, Taiwan
Sampling Method: Non-Probability Sample
Dates: Start 2008-08; Primary Completion 2008-10 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Ming Hsu,, M.D., Ph.D., Study Director — National Taiwan University Hospital